CLINICAL TRIAL: NCT06568471
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Clinical Study to Evaluate the Efficacy and Safety of HST101 in Chinese Patients with Hypercholesterolemia
Brief Title: A Study on Efficacy and Safety of HST101 in Chinese Patients with Hypercholesterolemia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hasten Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HST101-301
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Hypercholesterolemia; Dyslipidemias; Primary Hypercholesterolemia; Heterozygous Familial Hypercholesterolemia; Hyperlipidemia; Mixed; Metabolic Disease; ASCVD
Keywords: PCSK9 inhibitor; Lerodalcibep; LDL-C
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias; Hyperlipoproteinemia Type II; Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: All participants will be in-parallel randomized in a 2:1 ratio to HST101 or Placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study consists of the preceding 12-week double-blind, placebo-controlled treatment period and the subsequent 40-week (incluing 36-week HST101 treatment and 4-week follow-up) open-label treatment period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HST101(Lerodalcibep) (Experimental): 300 mg subcutaneously Q4W
  Interventions: Drug: Lerodalcibep
- Placebo (Placebo Comparator): subcutaneously Q4W
  Interventions: Drug: matching placebo

INTERVENTIONS:
Drug: Lerodalcibep — PCSK9 inhibitor
  Other Names: HST101; LIB003
  Arms: HST101(Lerodalcibep)
Drug: matching placebo — placebo
  Arms: Placebo

SUMMARY:
This randomized study is to assess LDL-C reductions at Week 12 with monthly (Q4W [≤31 days]) dosing of HST101 (lerodalcibep) 300 mg administered subcutaneously (SC) compared to placebo in patients with atherosclerotic cardiovascular disease (ASCVD) or very-high/high risk for ASCVD including Heterozygous familial hypercholesterolemia (HeFH) on a stable diet and oral LDL-C lowering drug therapy, followed by 36-week open-label treatment with subsequent 4-week follow-up for total 52-week long-term safety and efficacy evaluation.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled Phase 3 study. Participants who fulfill the inclusion and exclusion criteria will be enrolled at up to 35 study sites in mainland China.

All eligible participants will be randomized in a 2:1 ratio to HST101 or placebo dosed subcutaneously (Q4W [≤31 days]) in the initial 12-week randomized double-blind treatment period. After 12-week treatment, all the participants will enter to the 36-week open-label treatment period where those who are on HST101 will continue to receive HST101 in the same dosing regimen as dosed in the randomized period, and those who are on placebo will be switched to HST101 300 mg (Q4W [≤31 days]) administered subcutaneously.

The total study duration will be up to 55 weeks which includes a up to 3-week Screening Period, 12-week randomized, double-blind, placebo-controlled treatment period, 36-week open-label treatment period, followed by a 4-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written and signed informed consent form prior to any study-specific procedure;
* Male or female participants ≥18 years of age at the screening visit;
* Body weight ≥ 40 kg and body mass index (BMI) ≥18 and ≤35 kg/m2;
* On a stable diet and lipid-lowering oral drugs (such as statins, ezetimibe or Hybutimibe, omega-3 compounds, fenofibrate, nicotinic acid, etc.) for at least 4 weeks prior to the first drug administration
* LDL-C≥1.8 mmol/L (70 mg/dL) and TG≤4.52 mmol/L (400 mg/dL) at screening for ASCVD patients or those at very (ultra)-high risk for ASCVD, including patients with HeFH; LDL-C ≥ 2.6 mmol/L (100 mg/dL) and TG ≤ 4.52 mmol/L (400 mg/dL) at screening for patients at high-risk for ASCVD including patients with HeFH;
* Patients on a PCSK9 mAb at a dose of 75 mg, 140 mg, or 150 mg Q2W must undergo a washout period of ≥6 weeks after the last dose; for those on 300 mg or 420 mg Q4W, the washout period is ≥10 weeks following last dose;
* Female of childbearing potential must have a negative pregnancy test at the last screening visit and consent to use highly effective contraceptives during the trial and 3 months after the last dose of investigational drug.

Exclusion Criteria:

* Documented history of homozygous familial hypercholesterolemia (HoFH);
* Estimated glomerular filtration rate (eGFR)<30 mL/min/1.73m2;
* Active liver disease or hepatic dysfunction, history of liver transplant, and/or ALT or AST >2.5 × ULN at screening;
* Poorly controlled thyroid disorder including hypothyroidism or hyperthyroidism;
* Poorly controlled Type 1 or Type 2 diabetes mellitus defined as fasting blood glucose ≥11.0 mmol/L (200 mg/dL) and glycosylated hemoglobin (HbA1c) ≥ 9%;
* Serious arrhythmia, MI, unstable angina pectoris, PCI, CABG, implantable cardioverter defibrillator, aortic valve surgery or stroke within 3 months prior to the first dose;
* Planned cardiac surgery or revascularization during the study period;
* New York Heart Association (NYHA) Class III-IV heart failure;
* Pregnant or lactating women;
* Poorly controlled hypertension (SBP≥160 mmHg or DBP≥100 mmHg in a sitting position)
* Unexplained creatine kinase (CK) > 5 x ULN (retested once is needed if suspected to be related to excessive exercise or abnormal activity);
* LDL apheresis or plasma exchange within 2 months prior to the first dose;
* HIV, Treponema pallidum, or HCV antibody test positive, or HBV-DNA >ULN at screening;
* History of prescription drug abuse, illicit drug use or alcohol abuse within 6 months prior to screening;
* History of any major drug allergy, including allergy to protein biologics;
* Participate another clinical trial within 30 days or less than 5 half-lifes (drug) before screening, whichever is longer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-11-16 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
LDL-C change compared to Placebo | 12 weeks
  Percent change in LDL-C level from baseline (calculated by Friedewald formula) compared to Placebo
Mean LDL-C change at Weeks 10 and 12 compared to Placebo | 12 weeks
  Percent change in mean LDL-C level from baseline (calculated by Friedewald formula) compared to placebo at Weeks 10 and 12

SECONDARY OUTCOMES:
LDL-C change over time | 12 weeks
  Absolute and percent change in LDL-C level from baseline at Weeks 4, 8, 10, and 12
Free PCSK9 change | 12 weeks
  Absolute and Percent change in serum free PCSK9 level from baseline at Weeks 4,8 and 12
Other Lipid parameters change | 12 weeks
  Absolute and Percent change in TC, TG, HDL-C, non-HDL-C, VLDL-C, Apo B and Lp(a) from baseline at Weeks 4,8 and 12
Percentage of patients achieving LDL-C goals recommended by 2023 Chinese guideline | 12 weeks
  To assess the effect of HST101 on the percentage of patients achieving LDL-C<2.6 mmol/L (high-risk for ASCVD patients), LDL-C<1.8 mmol/L and >50% reduction from baseline (very-high risk for ASCVD patients), LDL-C<1.4 mmol/L and >50% reduction from baseline (ultra-high risk for ASCVD patients)
Incidence of treatment-emergent adverse events | 52 weeks
  Evaluation of adverse events, clinical lab tests, 12-lead ECG, vital signs, injection site reactions (ISRs)

OTHER OUTCOMES:
Long time free PCSK9 change | 52 weeks
  Absolute and percent change in serum free PCSK9 levels from baseline at Weeks 16,20,24,36,48 and 52
Long time LDL-C change | 52 weeks
  Absolute and percent change in LDL-C level from baseline at Weeks 16,20,22,24,36,48,50 and 52
Percentage of patients achieving LDL-C goals recommended by 2023 Chinese guideline | 52 weeks
  To assess the effect of HST101 on the percentage of patients achieving LDL-C<2.6 mmol/L (high-risk for ASCVD patients), LDL-C<1.8 mmol/L and >50% reduction from baseline (very-high risk for ASCVD patients), LDL-C<1.4 mmol/L and >50% reduction from baseline (ultra-high risk for ASCVD patients) at Weeks 16, 20, 24, 36, 48 and 52

CONTACTS AND LOCATIONS:
Overall Officials: Yong Huo, Principal Investigator — Peking University First Hospital
Locations (18):
- China (18):
  - Beijing Anzhen Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Beijing Luhe Hospital, Capital Medical Univeristy, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgeng Hospital, Beijing, Beijing Municipality
  - Fuwai Hospital, CAMS & PUMC, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Shijiazhuang People's Hospital, Shijiazhuang, Hebei
  - Daqingshi People's Hospital, Daqing, Heilingjiang
  - The 2nd Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanchang People's Hospital, Nanchang, Jiangxi
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Heze Municipal Hospital, Heze, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Zibo Municipal Hospital, Zibo, Shandong
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Wenzhou Medical Univesity, Wenzhou, Zhejiang
  - Peking University First Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No